CLINICAL TRIAL: NCT01459939
Title: A Double-blind, Randomized, Parallel Group, Fase III Comparative Study With Rose Hip Powder Powder and Placebo Given to Patients With Mild to Moderate Osteoarthritis in the Knee or/and Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hyben Vital ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HV 01/11
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Pain; Activities of Daily Living; Quality of Life
Keywords: Osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Daily treatment with placebo
  Interventions: Dietary Supplement: Placebo
- Rose-hip powder (Active Comparator): Daily treatment with Rose-hip powder
  Interventions: Dietary Supplement: Rose-hip powder capsules

INTERVENTIONS:
Dietary Supplement: Rose-hip powder capsules — 5 x 0,5 g rose-hip powder capsules BID the first 3 weeks and decreasing to 5 x 0,5 g QD the following 9 weeks
  Arms: Rose-hip powder
Dietary Supplement: Placebo — 5 x 0,5 g placebo powder capsules BID the first 3 weeks and decreasing to 5 x 0,5 g QD the following 9 weeks
  Arms: Placebo

SUMMARY:
The trial is an investigator-initiated, double-blind, randomized, placebo-controlled phase III study.

After the patient has receiving information about the study and after given written informed consent, the patient will be screened. All patients are randomized to receive standardized rose hip powder or matching placebo for 3 weeks followed by half the dose standardized rose hip (or placebo) for the remaining 12 weeks of the study.

The patient's medical history and demographic information will be recorded. The patient will then be asked questions in accordance to the study questionnaires, and they will also be asked to complete questionnaires regarding quality of life - and finally they be instructed on how to complete the diary.

Investigator or study nurse will take telephone contact with the subject after 3 and 6 weeks of treatment, subjects will be asked about how things are going and to remember to take the capsules and whether they have completed the diary.

The contact taken after 6 weeks by phone is mainly to guide the subject on how complete the questionnaires including VAS scales.

The last patient visit will take place after 12 weeks. Any side effects will be reported to and reviewed with HybenVital ApS in collaboration with medical experts.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 + years
* Osteoarthritis symptoms with duration of more than 6 months
* One WOMAC-pain visual analogue scale score (VAS score) there are at least 35 mm at rest
* Subjective morning joint stiffness
* Clinical symptoms of arthritis diagnosed by the ACR (American College Rheumatology) criteria

Exclusion Criteria:

* Patients who have been treated with rose hip extracts or powder within 3 months before screening.
* Patients who have been treated with ginger, avocado or soybean extracts or powder within 3 months before screening
* Patients on steroids, TNFalpha or DMARD prior to trial.
* Patients receiving irregular medical treatment for osteoarthritis.
* Patients suffering from other joint diseases other than osteoarthritis.
* Patients who abuse alcohol
* Patients with a current psychiatric illness, drug and / or alcohol abuse
* Patients with known allergy to rose hips
* Presence of other clinically significant medical conditions
* Patients scheduled for joint or major surgery during the trial.
* Patients participating in another clinical trial, or have participated in another clinical trial within 3 months before this study.
* Patients with known compliance problems or who are uncooperative.
* Pregnant or lactating women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
difference in the effect by using WOMAC-pain score. | 12 weeks
  The effect of treatment within each of the two groups (Rose hip powder and placebo) measured by using the differences in WOMAC-pain scores at 3 months of treatment between active treatment and placebo group, and between baseline and 3 months.
difference in the effect by using WOMAC-ADL score | 12 weeks
  The effect of treatment within each of the two groups (Rose hip powder and placebo) measured by using the differences in WOMAC-ADL (Activities of Daily Living) scores at 3 months of treatment between active treatment and placebo group, and between baseline and 3 months.

SECONDARY OUTCOMES:
Quality of life | 12 weeks
  Effects on QoL (SF-12 questionnaire and diaries) after 6 weeks and 12 weeks treatment, both groups compared to baseline, and the effects in the active group compared with the placebo group on QoL (SF-12 questionnaire and diaries) after 6 weeks and 12 weeks treatment.
Difference in the effect by using WOMAC-pain score | 6 weeks
  The effect of treatment within each of the two groups (Rose hip powder and placebo) measured by using the differences in WOMAC-pain scores at 6 weeks of treatment by compaing baseline to week 6, and the effects in the active group compared with the placebo group at 6 weeks
Patient assessment of the disease | 12 weeks
  Patient's assessment of the severity of the disease state is (PGAD)after 6 weeks and 12 weeks compareded to baseline and the effects in the active group compared with the placebo group at 6 and 12 weeks treatment
  Safety Issue?: (FDAAA) No
difference in the effect by using WOMAC-ADL (Activities of Daily Living)score | 6 weeks
  The effect of treatment within each of the two groups (Rose hip powder and placebo) measured by using the differences in WOMAC-ADL scores at 6 weeks of treatment by compaing baseline to week 6, and the effects in the active group compared with the placebo group at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pedersen, Dr, Principal Investigator — Aarhus University Hospital
Locations (1):
- INCUBA Science Park - Skejby, Aarhus, Denmark

REFERENCES:
- [Derived] Motawei AM, Warholm KM, Winther K. Using Dose-Response Correlation Re-Analyzing to Distinguish Placebo from Standardized Rose-Hip Powder (Lito) in a Clinical Trial on Osteoarthritis Where Data Initially Looked Identical. Nutrients. 2026 Jan 20;18(2):331. doi: 10.3390/nu18020331. PMID 41599942